CLINICAL TRIAL: NCT05590000
Title: Study of Gemini Rechargeable Spinal Cord Stimulation System
Brief Title: Study of Gemini Rechargeable Spinal Cord Stimulation (SCS) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ABT-CIP-10407
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Results first posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain
Keywords: Gemini rechargeable SCS System; ABT-CIP-10407; IPG
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Gemini rechargeable Spinal Cord Stimulation (SCS) System (Experimental): Patients will be implanted with the Gemini rechargeable SCS System
  Interventions: Device: Gemini SCS neuromodulation system

INTERVENTIONS:
Device: Gemini SCS neuromodulation system — This neurostimulation system is indicated as an aid in the management of chronic, intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with the following: failed back surgery syndrome, intractable low back and leg pain, angina pectoris and peripheral vascular disease.

SUMMARY:
The aim of this pre-market, prospective, single-arm, non-randomized, open-label, multi-center clinical study is to collect confirmatory data to show that the Gemini SCS neurostimulation system functions as intended in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is indicated for an SCS system, or has an implanted SCS system and is scheduled to receive an IPG replacement.
2. Subject is scheduled to receive a new IPG permanent implant and has completed a successful SCS trial in the last 6-months, OR subject is scheduled to undergo an all-in-one procedure OR has an implanted SCS system for an approved chronic pain indication.
3. Subject has a documented NRS pain score of ≥ 6 after at least 5 days without stimulation OR has an implanted functioning SCS system with NRS pain score of ≤ 4.
4. Subject must provide written informed consent prior to any clinical investigation-related procedure.
5. Subject is at least 18 years at the time of enrollment.
6. Subject is capable and willing to recharge an implanted IPG.

Exclusion Criteria:

1. Subject's SCS trial was unsuccessful.
2. Subject is currently participating, or intends to participate, in another clinical investigation that may confound the results of this study, as determined by Abbott.
3. Subject has or will receive more than one IPG.
4. Subject is pregnant or breastfeeding or plans to become pregnant during the clinical investigation follow-up period.
5. Subject has other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's assessment, could limit the subject's ability to participate in the clinical investigation.
6. Subject has or is scheduled to receive an intrathecal pump.
7. Subject is part of a vulnerable population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - QPain, Auchenflower
  - Metro Pain Group, Clayton
  - Sydney Spine & Pain, Hurstville
  - Sydney Pain Management Centre, Parramatta
  - Pain Care Perth, Perth
  - PainMedSA-Pain & Rehabilitation Specialists, Wayville

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled a total of 25 subjects at six investigational sites in Australia. The pre-market study enrolled the first subject on 20 September 2022 and the last subject on 09 December 2022. Completion of follow-up in the pre-market study occurred on 19 January 2023. One subject was withdrawn before IPG implantation without collection of baseline information. All other subjects were implanted and completed 2-week and 6-week visits.
Period: Overall Study
Arm/Group | Gemini Rechargeable Spinal Cord Stimulation (SCS) System
Started | 25
Completed | 24
Not Completed | 1
Not completed — The patient was indicated for peripheral nerve stimulation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemini Rechargeable Spinal Cord Stimulation (SCS) System
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 24
Primary Indication [Count of Participants; unit: Participants]
  Back Pain (No Prior Surgery) | 6
  Failed Back Surgery Syndrome - Fusion | 6
  Failed Back Surgery Syndrome - Non-Fusion | 3
  Reflex Sympathetic Dystrophy (Complex Regional Pain Syndrome Type I) | 2
  Other | 7
Time since chronic pain onset [Mean (Standard Deviation); unit: years] | 15.9 (13.4)
Manual therapy used to treat current condition [Count of Participants; unit: Participants]
  Yes | 21
  No | 3
Type of manual therapy used [Count of Participants; unit: Participants] — Population: 21 out of 24 implanted subjects received manual therapy prior to enrollment in the study.
  Participants
    Physical Therapy: number analyzed (Participants) | 21
    Physical Therapy | 21
    Occupational Therapy: number analyzed (Participants) | 21
    Occupational Therapy | 9
    Massage Therapy: number analyzed (Participants) | 21
    Massage Therapy | 10
    Chiropractic Therapy: number analyzed (Participants) | 21
    Chiropractic Therapy | 7
    Acupuncture: number analyzed (Participants) | 21
    Acupuncture | 1
Injections or interventions to treat current condition [Count of Participants; unit: Participants]
  Yes | 20
  No | 3
  Unknown | 1
Type of injection or intervention used [Count of Participants; unit: Participants] — Population: 20 out of 24 implanted subjects received injection or intervention prior to enrollment in the study
  Participants
    Epidural steroid injection: number analyzed (Participants) | 20
    Epidural steroid injection | 10
    Transforaminal: number analyzed (Participants) | 20
    Transforaminal | 7
    Translaminar: number analyzed (Participants) | 20
    Translaminar | 0
    Caudal: number analyzed (Participants) | 20
    Caudal | 5
    Facet joint injection: number analyzed (Participants) | 20
    Facet joint injection | 11
    Sacroiliac joint injection: number analyzed (Participants) | 20
    Sacroiliac joint injection | 5
    Radiofrequency ablation/rhizotomy: number analyzed (Participants) | 20
    Radiofrequency ablation/rhizotomy | 13
    Intradiscal therapy: number analyzed (Participants) | 20
    Intradiscal therapy | 0
    Intrathecal Pump: number analyzed (Participants) | 20
    Intrathecal Pump | 0

OUTCOME MEASURES:

1. Primary Outcome: Confirmatory Safety Endpoint: The Rate of Serious Adverse Events Related to the Investigational IPG and/or Charging System
Description: The rate of serious adverse events adjudicated as related to the investigational IPG and/or charging system will be assessed.
Time Frame: At 6 weeks (30-45 days) follow-up post implant
Population: ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemini Rechargeable Spinal Cord Stimulation (SCS) System
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 weeks after the permanent implant procedure
Arm/Group | Gemini Rechargeable Spinal Cord Stimulation (SCS) System
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemini Rechargeable Spinal Cord Stimulation (SCS) System (N=24)
CEREBROSPINAL FLUID LEAKAGE (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish the study results until publication of the results of the multi-center study or 2 years after study completion, whichever is sooner and allows the Sponsor to review any proposed publication at least 40 days before forwarding it to any person that is not bound by the confidentiality agreement between Sponsor and PI.

DOCUMENTS (2):
  • Study Protocol (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT05590000/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT05590000/SAP_001.pdf